CLINICAL TRIAL: NCT01353118
Title: Investigation of the Effects of Glycaemic Optimisation Before Gastric Bypass Surgery on the Glycaemic Remission and Microvascular Complication Rates of Type 2 Diabetes Mellitus
Brief Title: The Effects of Glycemic Optimization Before Gastric Bypass Surgery
Acronym: GLUCOSURG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Consultant metabolic medicine, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLUCOSURG 2
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; bariatric surgery; Roux-en-y gastric bypass; retinopathy; neuropathy; nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Retinal Diseases; Kidney Diseases | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gastric bypass (No Intervention): Group A: Patients will undergo gastric bypass surgery within 3 months after randomisation without any pre operative optimisation of glycaemic control.
- Gastric bypass 2 (Active Comparator): Gastric bypass 2 (Group B):Patients will undergo gastric bypass 3-6 months after randomisation. During this period the group will receive modern best medical care based on the American Diabetes Association (ADA)/European Association for the Study of Diabetes (EASD) guidelines. Glycaemic optimisation will be achieved in a gradual manner with particular attention to the avoidance of hypoglycaemia
  Interventions: Biological: gastric bypass

INTERVENTIONS:
Biological: gastric bypass — Optimise glucose control within 3 months before operation
  Other Names: Type 2 diabetes; glucose optimisation; microvascular complications; retinopathy; neuropathy; nephropathy; Gastric bypass with
  Arms: Gastric bypass 2

SUMMARY:
Metabolic surgery such as gastric bypass, gastric banding or sleeve gastrectomy operations can cause rapid and uncontrolled reductions in blood glucose. There is limited information on whether:

* metabolic surgery is superior to modern medical care for glycaemic control and type 2 diabetes remission.
* metabolic surgery is safe for microvascular complications of Type 2 diabetes
* good glycaemic control pre surgery has any effects on the long term glycaemia and complications of type 2 diabetes.

This study aims to assess:

1. whether metabolic surgery is better for diabetes control compared to medical treatment.
2. whether metabolic surgery is safe for eye, nerve and kidney complications.
3. whether good sugar control before metabolic surgery improves the long term effects of sugar control and microvascular complications.

DETAILED DESCRIPTION:
This is a prospective study involving 150 patients with type 2 diabetes mellitus (T2DM) and obesity. One hundred patients will undergo gastric bypass surgery whilst 50 will be treated with best medical care. The surgical patient group will be randomised to either immediate surgery or 3 months of medical glycaemic optimisation followed by surgery (n=50 group).

Intervention Group A: Patients will undergo gastric bypass surgery within 3 months after randomisation without any pre operative optimisation of glycaemic control.

Group B: Patients will undergo gastric bypass 3-6 months after randomisation. During this period the group will receive modern best medical care based on the American Diabetes Association (ADA)/European Association for the Study of Diabetes (EASD) guidelines. Glycaemic optimisation will be achieved with particular attention to the avoidance of hypoglycaemia.

Group C: Obese patients with T2DM (who choose not to have surgery) will be treated with best medical care based on the ADA/EASD guidelines including anti-diabetes/obesity pharmacotherapy, access to a trained dietician and exercise programme.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with T2DM and BMI above 35kg/m2
2. HbA1c ≥ 8.5% and/or the presence of at least one microvascular complication.

Exclusion Criteria:

* End stage retinopathy, nephropathy or neuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel Le Roux, MBChB, PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial Weight Centre, Charing Cross Hospital,, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gastric Bypass | Gastric Bypass 2
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No different
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Bypass | Gastric Bypass 2 | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 49 (5) | 48.5 (6) | 48.75 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
HbA1C [Mean (Standard Deviation); unit: %] | 10.3 (1.2) | 9.9 (1.1) | 10.1 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Fasting Glucose, Glycosylated Haemoglobin c and Rates of Type 2 Diabetes Mellitus Remission.
Description: A patient is considered to have achieved remission of T2F according to the American Diabetes Association criteria if they have fasting glucose below 6mmol/L AND HbA1c below 6% AND no medication for diabetes. Thus, a patient needs to achieve all of the three criteria (fasting glucose, HbA1C, and no medication) before being considered to be in remission. If a patient only achieves 2 of the criteria (fasting glucose and no medication) but the HbA1C is above 6% then they are not considered to be in remission.
  The outcome measure is calculated as the count of participants achiving the above criteria
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gastric Bypass | Gastric Bypass 2
Number analyzed (Participants) | 21 | 20
Participants | 6 | 6

2. Secondary Outcome: A Composite of Microvascular Complications
Description: A composite of microvascular complications. Microvascular events will be defined as new or worsening nephropathy, retinopathy or neuropathy.
  The outcome measure is calculated as the count of participants developing any of the microvascular events.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gastric Bypass | Gastric Bypass 2
Number analyzed (Participants) | 21 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Not different
Arm/Group | Gastric Bypass | Gastric Bypass 2
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 2/21 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Bypass (N=21) | Gastric Bypass 2 (N=20)
Hypoglycaemia (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes